CLINICAL TRIAL: NCT05235464
Title: Dissecting the Impact of Dietary Protein on Macrophage MTOR Signaling and Atherosclerosis
Brief Title: High Protein Diet and Atherosclerosis
Acronym: HPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2097342
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard meal (Active Comparator)
  Interventions: Other: Standard meal
- High animal protein meal (Experimental)
  Interventions: Other: High animal protein meal
- High plant protein meal (Experimental)
  Interventions: Other: High plant protein meal
- High plant protein meal with additional leucine (Experimental)
  Interventions: Other: High plant protein meal with additional leucine

INTERVENTIONS:
Other: Standard meal — Standard meal
  Arms: Standard meal
Other: High animal protein meal — Meal with high animal protein content
  Arms: High animal protein meal
Other: High plant protein meal — Meal with high plant protein content
  Arms: High plant protein meal
Other: High plant protein meal with additional leucine — Meal with high plant protein content and additional leucine
  Arms: High plant protein meal with additional leucine

SUMMARY:
Atherosclerosis is the underlying cause of the majority of cardiovascular diseases, including myocardial infarction and strokes, and results in tremendous morbidity and mortality. A Western-type diet is a major risk factor for atherosclerosis because of the high saturated fat, cholesterol, and refined carbohydrate contents. Dietary strategies to reduce cardiovascular disease burden therefore focus on restriction of saturated fat, cholesterol, and refined carbohydrates whereas "lean" protein intake is recommended and has become popular. However, results from studies conducted in animal models suggest high dietary protein intake is also atherogenic. The investigators' extensive preliminary data in animal models show that dietary protein increases atherosclerotic plaque formation and size and promotes necrotic core formation, a characteristic of rupture-prone plaques. The goal of the current proposal is to provide deeper insights into the relationship between protein intake and the pathogenesis of atherosclerosis by studying the mechanisms involved in protein-mediated atherogenesis and formation of necrotic plaques. The overarching hypothesis is that high protein intake drives atherosclerosis via leucine-mediated mTORC1 signaling in macrophages, which inhibits macrophage mitophagy and aggrephagy and stimulates macrophage proliferation. Furthermore, the investigators hypothesize that proteins from animal sources are more atherogenic than proteins from plant sources, because animal proteins contain more leucine than plant proteins. The investigators will test these hypotheses by using a sophisticated array of experimental strategies, including assays in primary macrophages and human monocyte-derived macrophages and genetically engineered mouse models. In addition, they will begin to translate the results obtained in vitro and in animals to people, and explore approaches to pharmacologically target the pro-atherogenic pathways as novel cardiovascular therapeutics. This proposal represents a paradigm shift in how a Western-type diet affects vascular health which has important implications since many adults in Western societies consume excess protein and dietary protein is heavily marketed for its presumed beneficial health effects.

ELIGIBILITY:
Inclusion Criteria:

* >=45 and <=75 years of age
* body mass index >=25.0 and <40.0 kg/m2

Exclusion Criteria:

* <45 and >75 years of age
* body mass index <25.0 or >39.9 kg/m2
* plasma triglyceride <125 mg/dl
* history of or current significant organ system dysfunction
* allergies or intolerances to meal ingredients
* use of medications or dietary supplements that could confound the study outcomes
* engaged in regular structured exercise >150 min per week
* alcohol use disorder
* premenopausal women
* persons who smoke
* prisoners
* inability to grant voluntary informed consent

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Monocyte p-S6 content | change from at 1 hour before meal intake and 3 hours after the meal
  phospho-S6 content in monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No